CLINICAL TRIAL: NCT00035607
Title: A Randomized, Open-label, Multicenter Study of Subcutaneous and Intravenous Administration of Darbepoetin Alfa (Novel Erythropoiesis Stimulating Protein, NESP) for the Treatment of Anemia in Subjects With Non-myeloid Malignancies Receiving Multicycle Chemotherapy
Brief Title: Chemotherapy Related Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20010199
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Anemia; Non-Myeloid Malignancies
MeSH Terms: conditions — Anemia

ARMS (2):
- Darbepoetin alfa SC (Active Comparator)
  Interventions: Drug: Darbepoetin alfa SC
- Darbepoetin alfa IV (Experimental)
  Interventions: Drug: Darbepoetin alfa IV

INTERVENTIONS:
Drug: Darbepoetin alfa SC — Subcutaneous (SC) injection of darbepoetin alfa at 4.5 mcg/kg weekly for weeks 1-6, then 4.5 mcg/kg Q3W
  Arms: Darbepoetin alfa SC
Drug: Darbepoetin alfa IV — Intravenous administration of darbepoetin alfa at 4.5 mcg/kg weekly for weeks 1-6, then 4.5 mcg/kg Q3W
  Arms: Darbepoetin alfa IV

SUMMARY:
This study is investigating darbepoetin alfa for the treatment of anemia in patients with non-myeloid cancers who are receiving chemotherapy. Darbepoetin alfa is a recombinant protein that stimulates the production of red blood cells. In this study, darbepoetin alfa will be administered as either an injection under the skin (subcutaneously) or directly into a vein (intravenously).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a non-myeloid malignancy
* Scheduled to receive a minimum of an additional 12 weeks of chemotherapy from the time of first dose of study drug
* Screening hemoglobin concentration less than or equal to 11.0g/dL
* ECOG performance status of 0 to 2
* Adequate renal and liver function

Exclusion Criteria:

* History of seizure disorder
* Received recombinant human erythropoietin (rHuEPO) or darbepoetin alfa therapy within 4 weeks before study day 1
* More than 2 red blood cell transfusions within 4 weeks before study day 1, or any red blood cell transfusion within 14 days before study day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-12; Primary Completion 2002-12 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration measured from baseline to the end of treatment period (EOTP) | from baseline to the end of treatment period (EOTP)

SECONDARY OUTCOMES:
Percentage of subjects who have a rapid rise in hemoglobin concentration; negative clinical consequences potentially associated with this rise evaluated in subjects with and without a rapid rise in hemoglobin concentration | throughout study
Change in hemoglobin concentration measured from baseline to week 7 and from week 7 to EOTP | from baseline to week 7 and from week 7 to EOTP
Time to and percentage of subjects who achieve hemoglobin improvement during the treatment period | during the treatment period
Time to and percentage of subjects with a hemoglobin response during the treatment period | during the treatment period
Percentage of subjects who exceed the hemoglobin threshold | throughout study
Incidence of all adverse events, serious adverse events, and severe or life-threatening adverse events | throughout study
Incidence, if any, of neutralizing antibody formation to darbepoetin alfa | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Justice G, Kessler JF, Jadeja J, Campos L, Weick J, Chen CF, Heatherington AC, Amado RG. A randomized, multicenter study of subcutaneous and intravenous darbepoetin alfa for the treatment of chemotherapy-induced anemia. Ann Oncol. 2005 Jul;16(7):1192-8. doi: 10.1093/annonc/mdi218. Epub 2005 Apr 28. PMID 15860486
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20010199.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/